CLINICAL TRIAL: NCT02345447
Title: Efficacy and Safety of an Herbal-Based Medication vs. Placebo in Preventing Acute Otitis Media in Children at High Risk of Recurrence: A Placebo Controlled, Randomized, Double-blinded Parallel-Group Comparison for Superiority
Brief Title: Herbal-Based Medication vs. Placebo in Preventing Acute Otitis Media in Children at High Risk of Recurrence
Acronym: OTV_PRE_01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Axel Franz, Associate Professor, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OTV.PRE.01.A3
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Herbal-based Medication (Active Comparator): Trade Name of active comparator: Otovowen® Substances: Aconitum napellus Dil. D6; Capsicum annuum Dil. D4; Chamomilla recutita; Echinacea purpurea; Hydrargyrum bicyanatum Dil. D6; Hydrastis canadensis Dil. D4; Iodum Dil. D4; Natrium tetraboracicum Dil. D4; Sambucus nigra; Sanguinaria canadensis.
  Manufacturer: Weber & Weber, Inning/Ammersee Dose: Three times daily 7 drops Mode of Application: orally Duration of Treatment: at first signs of Upper respirtory tract infection until symptoms resolve (maximally 8 weeks of continuous application).
  Interventions: Drug: Herbal-based medication
- Placebo (Placebo Comparator): Placebo Substance: Aqueous ethanol solution non-distinguishable from verum. Manufacturer: Weber & Weber, Inning/Ammersee Dose: Three times daily 7 drops Mode of Application: orally Duration of Treatment: at first signs of URI until symptoms resolve (maximally 8 weeks of continuous application).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Herbal-based medication — Aconitum napellus, Capsicum annuum; Chamomilla recutita; Echinacea purpurea; Hydrargyrum bicyanatum; Hydrastis canadensis; Iodum; Natrium tetraboracicum; Sambucus nigra; Sanguinaria canadensis
  Other Names: Otovowen(R)
  Arms: Herbal-based Medication
Drug: Placebo — Aqueous ethanol solution non-distinguishable from verum
  Arms: Placebo

SUMMARY:
The purpose of this study is to study whether a herbal-based medication is superior to placebo for prevention of acute otitis media in pre-school children with upper respiratory tract infection.

DETAILED DESCRIPTION:
This is a prospective, controlled parallel-group comparison for superiority of Otovowen®.

Patient will be identified by screening of patient cards. Patients with recurrent AOM aged 12 to 59 months will be randomly assigned either to Otovowen® or placebo. Randomization will be stratified by age at enrolment (12-35 versus 36-59 months).

The observation period per subject will be 6 months. Data collection and documentation will be performed weekly via online diary by the parents/legal representative(s) and by the investigator via eCRF.

Patients will be seen by the doctor at baseline and at end of study. Unscheduled visits in case of AOM or severe URI or any other disease are initiated by the parents/legal representative(s).

Study medication will be sent to the patient/parents/legal representative(s) after randomization. and will be administered at first signs or symptoms of URI (e. g. elevated temperature, common cold, influenza, coughing, sore throat, hoarse voice, frequent sneezing, running or stuffy nose, sinusitis, fever, headache, etc.) until resolved (maximally 8 weeks of continuous application).

AOM will be diagnosed during unscheduled visits according to the criteria detailed in the study protocol. An AOM will be considered as resolved through confirmation by the investigator only.

Compliance will be assessed by weighing contents of bottles of IMPs.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least 3 episodes of acute otitis media (AOM) within 12 months prior to study inclusion as documented in their medical records. Diagnosis criteria for AOM see study protocol
* parental written consent

Exclusion Criteria:

* Ongoing acute otitis media or URI
* Current prophylaxis/treatment for URI or AOM
* Current use of phytotherapeutic and homeopathic agents with secretolytic, anti-inflammatory or immune enhancing properties
* Use of tympanostomy tubes
* Chronic tympanic membrane perforation (TMP)
* Palatine cleft
* Parents/legal representative(s) of children unable to follow study procedures, who have no internet access and are not willing to use an online diary on a weekly basis
* History of hypersensitivity to the investigational drug or to its ingredients.
* Systemic, severe as well as history of uncontrolled chronic disease or a concurrent clinically significant illness, or medical condition, which in the investigator's opinion, would contraindicate study participation or compliance with protocol mandated procedures.
* Simultaneous participation in another clinical trial or participation in any clinical trial involving an investigational medicinal product within 30 days prior to written informed consent for this trial.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of acute otitis media episodes diagnosed by a physician | within 6 months after enrolment per patient

SECONDARY OUTCOMES:
Total number of acute otitis media per treatment group | diagnosed in each patient within 6 months after enrolment
Number of unscheduled visits due to AOM | within 6 months after enrolment
Number of AOM treated with antibiotics | within 6 months after enrolment
Number of unscheduled visits due to URI | within 6 months after enrolment
Number of URI treated with antibiotics | within 6 months after enrolment
Number of days with URI | within 6 months after enrolment
Subjective evaluation of efficacy by parent | at indivdual study completion 6 months after enrolment
Subjective evaluation of tolerability by parent | at indivdual study completion 6 months after enrolment
Occurence of adverse events | within 6 months of enrolment
number of days with use of antipyretic, analgesic and antibiotic medication | within 6 months of enrolment
Number of absent days from daycare (patient) / work (parent) | within 6 months of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Children's Hospital Tuebingen, Tübingen, Germany